CLINICAL TRIAL: NCT01538173
Title: Prospective Study Investigating the Role of Increased Microcirculation for Preventing Postoperative Surgical Side Infections in Patients Undergoing Reduction Mammoplasty
Brief Title: Increased Microcirculation for Preventing Postoperative Wound Infections in Patients Undergoing Reduction Mammoplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Max Dieterich (Other)
Collaborators: University of Rostock (Other)
Responsible Party: Sponsor-Investigator, Max Dieterich, Principle investigator, University of Rostock
Organization: University of Rostock (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BR02
Record Dates: First submitted 2012-02-19; First posted 2012-02-23 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Surgical Side Infections After Breast Reduction
Keywords: surgical side infection; breast reduction; reduction mammaplasty; prospective trial; microcirculation; breast surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HES group (Experimental): Application of twice a day 250ml HES 6% for three days postoperatively.
  Interventions: Drug: 250ml HES 6%
- NaCl group (Active Comparator): Application twice a day 500ml 9% NaCl for three days postoperatively.
  Interventions: Drug: 9% NaCl 500ml

INTERVENTIONS:
Drug: 250ml HES 6% — Application twice a day 250ml HES 6% for three days postoperatively.
  Arms: HES group
Drug: 9% NaCl 500ml — Application twice a day 500ml 9% NaCl for three days postoperatively.
  Arms: NaCl group

SUMMARY:
In this prospective study we investigated the impact of an improved postoperative microcirculation and its effect of surgical side infections after breast reduction.

DETAILED DESCRIPTION:
Many studies identifying risk factors for surgical side infections (SSI) after breast surgery included a large percentage of breast conserving therapies and risk factors for patients undergoing more extensive procedures like breast reduction (BR) are underrepresented and risk factors for more extensive breast surgeries might not be identified. Our approach to decrease SSI after BR was the application of an i.v. isotonic crystalloid solution, 6% hydroxyethylstaerke (HES) as a diminished peripheral blood flow and impaired vasculogenesis are characteristics of poorly healing wounds. HES causes a medium- to long-term increase in blood volume, blood flow and improved blood oxygen transport. Blood flow and tissue oxygenation are parts of regulating the healing process by utilizing molecular oxygen as a terminal oxidant. This antioxidant capacity can influence the wound healing process positively, as a characteristic feature of the inflammatory phase is the oxidative burst. HES additionally decreases haematocrite, blood viscosity and aggregation of erythrocytes positively influencing the complex components regulating wound healing. These characteristics and the increase in blood circulation might influence the postoperative healing and regeneration process.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients were at least 18 years of age, scheduled for breast reduction, guaranteed follow-up of 30 days.

Exclusion Criteria:

* Patients were excluded if they had a history of coagulopathy or history of antiplatelet agent use within 10 days of surgery

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Actual)
Dates: Start 2007-01; Primary Completion 2011-10 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Surgical side infection | 4 weeks
  Primary end point was the development of surgical side infection

SECONDARY OUTCOMES:
Risk factors | 4 weeks
  Secondary endpoints were identification of possible risk factors for surgical side infections and nipple necrosis after breast reduction.

CONTACTS AND LOCATIONS:
Overall Officials: Max Dieterich, MD, Principal Investigator — University of Rostock
Locations (1):
- University of Rostock, Department of Obstetrics and Gynecology, Rostock, Mecklenburg-Vorpommern, Germany